CLINICAL TRIAL: NCT05405374
Title: A Prospective, Randomized, Intra-Patient Controlled, Multi-Center Clinical Investigation Evaluating OSTEOAMP SELECT Fibers Versus Infuse Bone Graft as Autograft Substitute in Lumbar Fusion Procedures
Brief Title: OSTEOAMP Lumbar Fusion Intra-Patient Controlled Study
Acronym: SELECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bioventus LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGS-21-01
Record Dates: First submitted 2021-12-09; First posted 2022-06-06 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Lumbar Spine Disease; Lumbar Spondylolisthesis; Lumbar Spine Instability; Lumbar Spondylosis; Degenerative Disc Disease
Keywords: Lumbar Interbody Fusion
MeSH Terms: conditions — Spinal Diseases; Spondylolisthesis; Spondylosis; Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: In this study, all subjects will be treated at 2 levels of the anterior lumbar spine. One of the levels will be grafted with OSTEOAMP SELECT and the other with Infuse housed within the same type of interbody cage. The assignment of the bone graft product to each treated motion segment will be randomized in a 1:1 ratio. Every subject will serve as his/her own control.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- OSTEOAMP (Active Comparator): OSTEOAMP SELECT Fibers as an autograft substitute in lumbar interbody fusion procedures
  Interventions: Other: OSTEOAMP
- Infuse (Active Comparator): The Infuse Bone Graft as an autograft substitute in lumbar interbody fusion procedures
  Interventions: Device: Infuse

INTERVENTIONS:
Other: OSTEOAMP — OSTEOAMP SELECT Fibers (derived from human bone allograft) rehydrated with bone marrow aspirate (BMA) and combined with local autogenous graft for use in lumbar interbody fusion of the lumbar spine.
  Arms: OSTEOAMP
Device: Infuse — The Infuse Bone Graft/Medtronic Interbody Fusion Device consists of recombinant human Bone Morphogenetic Protein-2 (rhBMP-2, known as dibotermin alfa) placed on an absorbable collagen sponge (ACS). rhBMP-2 is the active agent in the Infuse Bone Graft component. The ACS is a soft, white, pliable, absorbent implantable matrix for rhBMP-2.
  Arms: Infuse

SUMMARY:
The objective of this clinical study is to compare OSTEOAMP SELECT Fibers to Infuse Bone Graft, in terms of effectiveness and safety, when used as a bone graft substitute in in skeletally mature patients qualified for 2-lumbar interbody fusion (LIF) by means of an intra-patient control model.

DETAILED DESCRIPTION:
The current study will collect clinical evidence for OSTEOAMP SELECT in spinal fusion procedures. In particular, the study will explore the use of OSTEOAMP SELECT as part of a lumbar interbody fusion (LIF) procedure of two lumbar motion segments between L2 to S1 in patients suffering from symptomatic degenerative disc disease (DDD), degenerative spondylolisthesis, and/or mild degenerative scoliosis.

Effectiveness will be based on the lumbar interbody fusion rate at the index levels assessed by a treatment-blinded independent reviewer at 12 months and 24 months.

Safety will be evaluated by documenting the number and nature of all (serious) adverse events that may in any way be related to the surgical procedure or product. The complication rate will be compared to the rate in control populations from literature.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature male or female patient, at least 21 years of age and no more than 80 years of age, inclusive, at the time of surgery;
* Has symptomatic degenerative disc disease (DDD) of the lumbosacral spine in two levels (L2 to S1). Lumbar DDD is defined as discogenic back pain with or without radicular symptoms confirmed by patient history and radiographic studies
* Has radiographic evidence (e.g. CT, MRI, x-ray, etc.) of degenerative lumbosacral disease including instability up to and including Grade 1 spondylolisthesis at the involved level(s)
* Requires fusion (i.e., symptomatic) at 2 adjacent or non-adjacent levels from L2 to S1;
* Non-responsive to non-operative treatment (e.g., bed rest, physical therapy, medication,spinal injection, manipulation, and/or TENS) for at least 6 months;
* Willing and able to comply with the study protocol (including post-operative clinical and radiographic evaluations and required rehabilitation plan) and able to understand and sign the Informed Consent.

Exclusion Criteria:

* Previous lumbar spine surgery with the exception of discectomy and/or laminectomy at the target levels.
* Lumbar scoliosis >30 degrees.
* Documented history of osteoporosis, osteomalacia, Paget's disease or metabolic bone disease
* Morbidly obese, as defined by a Body Mass Index (BMI) >40 kg/m2.
* Documented history of uncontrolled diabetes mellitus
* Presence of active malignancy or prior history of malignancy (non-invasive basal cell carcinoma of the skin is allowed).
* Overt or active bacterial infection, either local to surgical space or systemic.
* Chronic use of steroids (defined as more than 6 weeks of steroid use within 12 months of surgery, other than episodic use or inhaled corticosteroids)
* Co-morbidities, which in the investigator's opinion, precludes the subject from being a surgical candidate.
* Autoimmune disease, which in the investigator's opinion, is known to affect bone metabolism or the spine (e.g., spondyloarthropathies, juvenile arthritis, rheumatoid arthritis, Graves' disease, Hashimoto's thyroiditis).
* Any endocrine or metabolic disorder, which in the investigator's opinion, is known to affect osteogenesis (e.g., Paget's disease, renal osteodystrophy, Ehlers- Danlos syndrome, or osteogenesis imperfecta).
* History of hypersensitivity and/or allergy to any of the agents used to process OSTEOAMP SELECT, including bacitracin, polymyxin B sulfate, and gentamicin.
* Known hypersensitivity or allergy to any components of the study treatments including, but not limited to bone morphogenetic proteins (BMPs); injectable collagen; protein pharmaceuticals (e.g., monoclonal antibodies or gamma globulins); bovine collagen products; and/or instrumentation materials (e.g., titanium, titanium alloy, cobalt chrome,cobalt chrome alloy, or PEEK).
* Is a prisoner.
* Treatment with an investigational therapy (drug, device, and/or biologic) targeting spinal conditions within 3 months prior to implantation surgery, treatment with any other investigational therapies within 30 days prior to implantation surgery, or such treatment is planned during the 24-month period following implantation of the study treatment.
* Pregnant or nursing. Females of child-bearing potential must agree not to become pregnant for the duration of the study.
* A history of alcohol and/or drug abuse within 6 months prior to screening or exhibits evidence, in the investigator's opinion, of alcohol/drug abuse at screening.
* Current history of heavy nicotine use (e.g. more than 20 cigarettes per day).
* Any condition, which in the investigator's opinion, would interfere with the subject's ability to comply with study instructions, which might confound data interpretation.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Fusion Status | 12 Months
  Radiographic fusion as defined by the Image Review Charter and assessed by an independent core laboratory.

SECONDARY OUTCOMES:
Fusion Status | 24 Months
  Radiographic fusion as defined by the Image Review Charter and assessed by an independent core laboratory.

OTHER OUTCOMES:
Functional Impairment | 24 Months
  Derived from the Oswestry Low Back Pain Questionnaire to quantify low back pain and function. Zero is equated with no disability and 100 is the maximum disability possible.
Back Pain | 24 Months
  Visual Analogue Scale (VAS) change in back pain from baseline to 24 month follow up assessed at time frames: Pre-Op, 6 weeks, 3 month, 6 month, 12 month, 24 month.
  Visual Analogue Scale is rated from 0 - 10 cm (no pain - worst possible pain)
Leg Pain | 24 Months
  Visual Analogue Scale (VAS) change in leg pain from baseline to 24 month follow up assessed at time frames: Pre-Op, 6 weeks, 3 month, 6 month, 12 month, 24 month.
  Visual Analogue Scale is rated from 0 - 10 cm (no pain - worst possible pain)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Yale University, New Haven, Connecticut
  - Kansas Joint and Spine Specialists, Wichita, Kansas
  - Orthopaedic Institute of Western Kentucky, Paducah, Kentucky
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - New England Baptist Hospital, Boston, Massachusetts
  - Tennessee Orthopaedic Alliance, Nashville, Tennessee
  - Austin Neurosurgeons, Austin, Texas
  - OrthoVirginia, Richmond, Virginia
  - West Virginia University, Morgantown, West Virginia